CLINICAL TRIAL: NCT06393400
Title: An Open-label, Single-arm, Phase 1 Study of the Combination of FMT and Gemcitabine with Nab-paclitaxel As First-line Therapy in Patients with Advanced Pancreatic Ductal Adenocarcinoma.
Brief Title: CHemotherapy and Stool Transplant in PDAC (CHASe-PDAC)
Acronym: CHASe-PDAC
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: John Lenehan (Other)
Responsible Party: Sponsor-Investigator, John Lenehan, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Organization: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ReDA 14577
Record Dates: First submitted 2024-04-18; First posted 2024-05-01 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Unresectable or Metastatic Advanced Pancreatic Ductal Adenocarcinoma
Keywords: PDAC, Fecal Microbial Transplantation, Gut Microbiome
MeSH Terms: conditions — Anophthalmia with pulmonary hypoplasia | interventions — Fecal Microbiota Transplantation; polyethylene glycol 3350; Gemcitabine; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Fecal Microbiota Transplantation (Experimental): A single Fecal Microbiota Transplantation (FMT) with 100 g of healthy stool in 36-40 oral capsules once 24 hours after Polyethylene Glycol laxative preparation, followed by gemcitabine 1000 mg/m2 intravenously (IV) and nab-paclitaxel 125 mg/m2 IV on Day 1, Day 8, and Day 15 of each 28-day cycle at least 7 days after FMT.
  Interventions: Drug: Fecal Microbiota Transplantation; Drug: PEG3350; Drug: Gemcitabine; Drug: nab-Paclitaxel

INTERVENTIONS:
Drug: Fecal Microbiota Transplantation — Fecal Microbiota Transplantation with 100 g of healthy donor stool in 36-40 oral capsules once
  Other Names:
  * FMT
  * Stool Transplant
  * Poop Transplant
Drug: PEG3350 — Polyethylene Glycol 3350 17 g oral dissolved in 4 litres of water consumed the evening before FMT.
  Other Names:
  * PEG3350
  * RestoraLAX
  * MiraLAX
Drug: Gemcitabine — Gemcitabine 1000 mg/m2/day IV on Days 1, 8, and 15 of each 28-day cycle.
  Other Names:
  - Gemzar
Drug: nab-Paclitaxel — nab-Paclitaxel 125 mg/m2/day IV on Days 1, 8, and 15 of each 28-day cycle.
  Other Names:
  - Abraxane

SUMMARY:
To confirm the safety of combining oral fecal microbiota transplantation (FMT) with gemcitabine and nab-paclitaxel chemotherapy as first line treatment in patients with unresectable or metastatic pancreatic ductal adenocarcinoma.

DETAILED DESCRIPTION:
This is a phase 1 open-labelled, non-randomized safety trial examining oral fecal microbiota transplantation (FMT) with healthy donor stool in combination with standard of care (SOC) gemcitabine and nab-paclitaxel (GnP) in patients with advanced (unresectable and metastatic) pancreatic ductal adenocarcinoma (PDAC) as first-line therapy. A total of 20 eligible patients will be treated with study treatment. The purpose of the trial is to confirm the safety of combined therapy, assess clinical outcomes, perform gut microbiome analysis, systemic immune profiling, and explore patient-related outcomes. This trial will be conducted at the Verspeeten Family Cancer Centre (formerly known as the London Regional Cancer Program) at London Health Sciences Centre.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be 18-years old or older
* Patients must have a confirmed diagnosis of unresectable or metastatic pancreatic ductal adenocarcinoma. Diagnosis confirmation may include pathologic assessment or radiographic/biomarker determination of PDAC when obtaining a tumour sample is not feasible/successful. The latter case requires review at the Pancreas Multi-disciplinary Case Conference (MCC)
* Patients with ECOG performance of 0-2
* Patients who have consented to treatment with first-line gemcitabine with nab-paclitaxel at the discretion of their primary oncologist. Patients must receive at least one dose of both chemotherapy agents to be considered eligible for evaluation.
* Patients must be able to provide written informed consent and understand the infectious risks associated with FMT administration
* Patients must understand that there are non-infectious risks associated with FMT administration
* Ability to ingest capsules
* Understand that data regarding the long-term safety risk of FMT are lacking
* Have evaluable disease as per RECIST version 1.1

Patients may receive other localized therapies with palliative intent while on therapy to include external beam radiation to areas of metastatic disease. Stratification of outcomes will include identifying patients that receive palliative radiation to the primary tumour itself.

Exclusion Criteria:

* Previously received cytotoxic chemotherapy with curative or non-curative intent for PDAC
* Pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit
* Has a diagnosis of immunodeficiency (e.g. HIV, organ transplantation)
* Ongoing use of antibiotics or previous use of antibiotics within 7 days prior to the FMT procedure
* Probiotic supplements and food products labeled as containing probiotics must be discontinued a minimum of 72 hours before FMT administration and are not permitted during the first 3 months of chemotherapy treatment
* Presence of a chronic intestinal disease (e.g. Celiac, malabsorption, primary colonic tumor)
* Presence of absolute contra-indications to FMT administration

  * Toxic megacolon
  * Severe dietary allergies (e.g. shellfish, nuts, seafood)
  * Inflammatory bowel disease
* Has serious concomitant illnesses, such as: cardiovascular disease (uncontrolled congestive heart failure, uncontrolled hypertension, cardiac ischemia, myocardial infarction, and severe cardiac arrhythmia), bleeding disorders, autoimmune diseases, severe obstructive or restrictive pulmonary diseases, active systemic infections, and inflammatory bowel disorders

  * This includes HIV or AIDS-related illness, or active HBV and HCV
* Has an active infection requiring systemic therapy
* Patient has received a live vaccine within 4 weeks prior to the first dose of treatment

  * Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial

Special considerations include patients who are unable to tolerate the combination of gemcitabine with nab-paclitaxel, and subsequently after starting chemotherapy are transitioned to gemcitabine alone at the discretion of their treating oncologist. Such patients will not be removed or disqualified from continuing in the study but their clinical outcomes will be stratified between those who received nab-paclitaxel with gemcitabine and those who transitioned to gemcitabine alone. In general, this scenario is not expected to commonly occur in this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-01-08 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | Approximately end of year 4 (Study Completion)
  FMT in combination with systemic therapy in patients with advanced PDAC has not been studied to our knowledge. Prior to proceeding with a larger study, this phase I study will include 20 patients receiving G-nP who will receive a single FMT with healthy donor stool prior to the first dose of chemotherapy. There are well-known toxicities associated with these 2 chemotherapeutic agents, several of which affect the gastrointestinal tract. The most common side effects resulting from FMT are primarily mild gastrointestinal effects. FMT has been found to be safe when combined with ICIs and there has been no increase in the number of toxicities or severity observed. The measure of safety in this trial will be assessing for treatment-related adverse events that will be graded according to the NCI-CTCAE v5. A positive trial result with respect to toxicity will be designated if there are no unexpected or more severe toxicities associated than with the chemotherapy drugs alone.

SECONDARY OUTCOMES:
Progression-Free Survival | Time between study enrollment and the time of disease progression, death, or date of last follow-up, whichever occurs first.
  Determined using RECIST 1.1 criteria to evaluate changes in tumour size on routine imaging and quantified using the Kaplan-Meier method.
Overall Survival | Until the date of death from any cause assessed from the date of FMT up to 24 months.
  Quantified using the Kaplan-Meier method alone.
Tolerability of consuming the FMT capsules | 24 months
  The tolerability of consuming approximately 40 capsules in patients with PDAC will be assessed by study personnel through direct observation of the FMT process. Patients with advanced PDAC are often unwell, cachectic, anorexic, and experiencing nausea associated with the cancer process. Adequate intake of calories and hydration are routinely a challenge in this patient population. Before a larger study can be contemplated, the feasibility and tolerability of consuming the large number of capsules needs to be demonstrated in a smaller study like this.
Objective Response Rate | Approximately 4 years (end of study)
  A reduction in size of PDAC tumours is often not achieved or dramatic when they occur, therefore the ORR is not considered a benchmark of success in this study. However, some patients may benefit from a reduction in tumour volume with respect to cancer-related symptoms such as gastric outlet obstruction resulting from extrinsic compression by the tumour. The ORR will be assessed given its potential to be clinically meaningful and will be determined using the RECIST 1.1 criteria.
Clinical Benefit Rate | Approximately 4 years (end of study)
  The CBR may be more clinically relevant to patients with PDAC where SD directly relates to the duration of PFS and few achieve a CR or PR.

CONTACTS AND LOCATIONS:
Locations (1):
- Verspeeten Family Cancer Centre (formerly known as the London Regional Cancer Program) London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No